CLINICAL TRIAL: NCT00663208
Title: Double-Blind, Placebo-Controlled, Multiple Ascending Dose Study to Evaluate the Antiviral Activity and Safety, Tolerability, and Pharmacokinetics of Daclatasvir in Subjects Infected With Hepatitis C Virus Genotype 1
Brief Title: A Multiple Ascending Dose Study of Daclatasvir (BMS-790052) in Hepatitis C Virus Genotype 1 Infected Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AI444-004
Record Dates: First submitted 2008-04-18; First posted 2008-04-22 (Estimated); Results first posted 2015-10-14 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-09

CONDITIONS: Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — daclatasvir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Group 1 (Active Comparator): Daclatasvir (1 mg), once daily
  or
  Matching Placebo, once daily
  Interventions: Drug: Daclatasvir; Drug: Placebo
- Group 2 (Active Comparator): Daclatasvir (10 mg), once daily
  or
  Matching Placebo, once daily
  Interventions: Drug: Daclatasvir; Drug: Placebo
- Group 3 (Active Comparator): Daclatasvir (1-100 mg), once or twice daily
  or
  Matching Placebo, once or twice daily
  Interventions: Drug: Daclatasvir; Drug: Placebo
- Group 4 (Active Comparator): Daclatasvir (1-100 mg), once or twice daily
  or
  Matching Placebo, once or twice daily
  Interventions: Drug: Daclatasvir; Drug: Placebo
- Group 5 (Active Comparator): Group 5: Active Comparator
  Daclatasvir (1-100 mg), once or twice daily
  or
  Matching Placebo, once or twice daily
  Interventions: Drug: Daclatasvir; Drug: Placebo
- Group 6 (Active Comparator): Group 6: Active Comparator
  Daclatasvir (1-100 mg), once or twice daily
  or
  Matching Placebo, once or twice daily
  Interventions: Drug: Daclatasvir; Drug: Placebo

INTERVENTIONS:
Drug: Daclatasvir — Capsule, Oral, Approximately 182 days from initial dosing
Drug: Placebo — Capsule, Oral, After 28 days from initial dosing and unblinding of the dose panel

SUMMARY:
The primary purpose of this study is to assess the change in Hepatitis C Virus RNA during dosing with daclatasvir and during the follow-up period in subjects with chronic hepatitis C infection

ELIGIBILITY:
Inclusion Criteria:

* Chronically infected with Hepatitis C Virus (HCV) genotype 1
* Treatment naive or treatment non-responders or treatment intolerant; and not co-infected with HIV or Hepatitis B Virus
* HCV RNA viral load of ≥10*5 IU/mL
* BMI 18 to 35kg/m²

Exclusion Criteria:

* Any significant acute or chronic medical illness which is not stable or is not controlled with medication and not consistent with Hepatitis C Virus infection
* HIV and/or HBV positive
* Major surgery within 4 weeks of study drug administration and any gastrointestinal surgery that could impact the absorption of study drug

WOCBP will be enrolled as in-patient for 16 days

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 167 (Actual)
Dates: Start 2008-05; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (8):
- United States (7):
  - Advanced Clinical Res Inst, Anaheim, California
  - West Coast Clinical Trials, Llc, Cypress, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Elite Research Institute, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - Parexel International Corporation, Baltimore, Maryland
  - Alamo Medical Research, San Antonio, Texas
- Local Institution, Santurce, Puerto Rico

REFERENCES:
- [Derived] Nettles RE, Gao M, Bifano M, Chung E, Persson A, Marbury TC, Goldwater R, DeMicco MP, Rodriguez-Torres M, Vutikullird A, Fuentes E, Lawitz E, Lopez-Talavera JC, Grasela DM. Multiple ascending dose study of BMS-790052, a nonstructural protein 5A replication complex inhibitor, in patients infected with hepatitis C virus genotype 1. Hepatology. 2011 Dec;54(6):1956-65. doi: 10.1002/hep.24609. PMID 21837752
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 167 enrolled; 30 entered treatment Period. Reasons for not entering: 1 lost to follow-up, 4 withdrew consent, 5 administrative reasons, 6 other, 121 did not meet study criteria.
Pre-assignment Details: A total of 30 participants received study treatment.
Groups:
- Daclatasvir (1 mg) QD: Participants received once daily (QD) dose of daclatasvir 1 mg during 14 day treatment period. Participants who received daclatasvir were followed up at Day 28, Day 42, Day 98 and Day 182.
- Daclatasvir (10 mg) QD: Participants received QD dose of daclatasvir 10 mg during 14 day treatment period. Participants who received daclatasvir were followed up at Day 28, Day 42, Day 98 and Day 182.
- Daclatasvir (30 mg) QD: Participants received QD dose of daclatasvir 30 mg during 14 day treatment period. Participants who received daclatasvir were followed up at Day 28, Day 42, Day 98 and Day 182.
- Daclatasvir (60 mg) QD: Participants received QD dose of daclatasvir 60 mg during 14 day treatment period. Participants who received daclatasvir were followed up at Day 28, Day 42, Day 98 and Day 182.
- Daclatasvir (30 mg) BID: Participants received twice daily (BID) dose of daclatasvir 30 mg during 14 day treatment period. Participants who received daclatasvir were followed up at Day 28, Day 42, Day 98 and Day 182.
- Daclatasvir (100 mg) QD: Participants received QD dose of daclatasvir 100 mg during 14 day treatment period. Participants who received daclatasvir were followed up at Day 28, Day 42, Day 98 and Day 182.
- Placebo: Participants received QD/BID dose of placebo matched to daclatasvir during 14 day treatment period. Participants who received placebo were discharged after Day 28 and after unblinding of the dose panel.
Period: Treatment Period
Arm/Group | Daclatasvir (1 mg) QD | Daclatasvir (10 mg) QD | Daclatasvir (30 mg) QD | Daclatasvir (60 mg) QD | Daclatasvir (30 mg) BID | Daclatasvir (100 mg) QD | Placebo
Started | 4 | 4 | 4 | 4 | 4 | 4 | 6
Completed | 4 | 3 | 4 | 4 | 4 | 4 | 6
Not Completed | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 0 | 0
Period: Follow-up Period
Arm/Group | Daclatasvir (1 mg) QD | Daclatasvir (10 mg) QD | Daclatasvir (30 mg) QD | Daclatasvir (60 mg) QD | Daclatasvir (30 mg) BID | Daclatasvir (100 mg) QD | Placebo
Started | 4 | 3 | 4 | 4 | 4 | 4 | 6
Completed | 1 | 3 | 1 | 2 | 4 | 4 | 5
Not Completed | 3 | 0 | 3 | 2 | 0 | 0 | 1
Not completed — Lost to Follow-up | 2 | 0 | 3 | 2 | 0 | 0 | 0
Not completed — Other reason | 1 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The analysis was performed on all treated participants.
Groups:
- Daclatasvir (1 mg) QD: Participants received QD dose of daclatasvir 1 mg during 14 day treatment period. Participants who received daclatasvir were followed up at Day 28, Day 42, Day 98 and Day 182.
- Daclatasvir (30 mg) BID: Participants received BID dose of daclatasvir 30 mg during 14 day treatment period. Participants who received daclatasvir were followed up at Day 28, Day 42, Day 98 and Day 182.
- Total: Total of all reporting groups
Arm/Group | Daclatasvir (1 mg) QD | Daclatasvir (10 mg) QD | Daclatasvir (30 mg) QD | Daclatasvir (60 mg) QD | Daclatasvir (30 mg) BID | Daclatasvir (100 mg) QD | Placebo | Total
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 6 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.5 (9.95) | 46.5 (13.00) | 47.5 (3.70) | 39.5 (7.55) | 44.8 (6.40) | 44.3 (6.90) | 48.0 (4.20) | 44.5 (7.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 5
  Male | 3 | 3 | 4 | 3 | 4 | 3 | 5 | 25

OUTCOME MEASURES:

1. Secondary Outcome: Change From Baseline at Day 7 in log10 Hepatitis C Virus (HCV) RNA Levels of Participants Without Baseline Drug Resistance
Description: The Roche TaqMan HCV quantitative assay was used for analysis with detection limit of 10 international units/ millilitre (IU/mL). Baseline was Day -1
Time Frame: Baseline, Day 7
Population: All randomized participants who took at least 1 dose of study medication.
Measure: Mean (90% Confidence Interval); unit: log10 IU/mL
Arm/Group | Daclatasvir (1 mg) QD | Daclatasvir (10 mg) QD | Daclatasvir (30 mg) QD | Daclatasvir (60 mg) QD | Daclatasvir (30 mg) BID | Daclatasvir (100 mg) QD | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 3 | 3 | 3 | 6
log10 IU/mL | -2.13 [-3.10 to -1.16] | -3.31 [-4.28 to -2.34] | -2.91 [-3.88 to -1.94] | -2.58 [-3.55 to -1.61] | -3.03 [-4.00 to -2.07] | -3.56 [-4.52 to -2.59] | 0.00 [-0.86 to 0.87]

2. Primary Outcome: Change From Baseline at Day 7 in log10 Hepatitis C Virus (HCV) RNA of All Participants
Description: The Roche TaqMan HCV quantitative assay was used for analysis with detection limit of 10 IU/mL. Baseline was Day -1.
Time Frame: Baseline, Day 7
Population: All randomized participants who took at least 1 dose of study medication.
Measure: Mean (90% Confidence Interval); unit: log10 IU/mL
Arm/Group | Daclatasvir (1 mg) QD | Daclatasvir (10 mg) QD | Daclatasvir (30 mg) QD | Daclatasvir (60 mg) QD | Daclatasvir (30 mg) BID | Daclatasvir (100 mg) QD | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 6
log10 IU/mL | -2.13 [-3.10 to -1.16] | -3.31 [-4.28 to -2.34] | -2.91 [-3.88 to -1.94] | -2.58 [-3.55 to -1.61] | -3.03 [-4.00 to -2.07] | -3.56 [-4.52 to -2.59] | 0.00 [-0.86 to 0.87]

3. Secondary Outcome: Change From Baseline at 24 h Post Dose on Day 1 in log10 Hepatitis C Virus (HCV) RNA of Participants Without Baseline Drug Resistance
Description: The Roche TaqMan HCV quantitative assay was used for analysis with detection limit of 10 IU/mL. Baseline was Day -1.
Time Frame: Baseline, 2, 4, 6, 8, 12, 16, 20, and 24 hours post dose on Day 1
Population: All randomized participants who took at least 1 dose of study medication and did not have baseline genotypic drug resistance mutations were summarized.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | Daclatasvir (1 mg) QD | Daclatasvir (10 mg) QD | Daclatasvir (30 mg) QD | Daclatasvir (60 mg) QD | Daclatasvir (30 mg) BID | Daclatasvir (100 mg) QD | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 3 | 3 | 3 | 6
log10 IU/mL
  Change at Hour 2 | 0.02 (0.137) | -0.00 (0.083) | -0.21 (0.244) | -0.43 (0.324) | -0.35 (0.284) | 0.04 (0.107) | -0.00 (0.216)
  Change at Hour 4 | -0.78 (0.273) | -0.91 (0.206) | -1.22 (0.202) | -1.24 (0.711) | -1.24 (0.397) | -1.01 (0.345) | 0.07 (0.248)
  Change at Hour 6 | -1.47 (0.466) | -1.73 (0.272) | -2.05 (0.237) | -1.96 (0.717) | -1.99 (0.552) | -1.36 (0.473) | 0.00 (0.209)
  Change at Hour 8 | -1.92 (0.516) | -2.12 (0.216) | -2.62 (0.195) | -2.47 (0.733) | -2.59 (0.509) | -1.74 (0.917) | -0.01 (0.251)
  Change at Hour 12 | -2.18 (0.439) | -2.44 (0.092) | -2.91 (0.083) | -3.08 (0.562) | -2.92 (0.511) | -2.00 (1.158) | -0.01 (0.284)
  Change at Hour 16 | -2.09 (0.420) | -2.76 (0.183) | -2.95 (0.250) | -3.38 (0.521) | -3.04 (0.535) | -2.03 (1.009) | -0.00 (0.246)
  Change at Hour 20 | -1.92 (0.447) | -2.80 (0.095) | -3.02 (0.086) | -3.50 (0.312) | -3.38 (0.477) | -2.29 (1.240) | 0.01 (0.155)
  Change at Hour 24 | -1.82 (0.480) | -2.97 (0.216) | -3.24 (0.103) | -3.60 (0.204) | -3.53 (0.624) | -2.58 (1.292) | 0.02 (0.246)

4. Secondary Outcome: Change From Baseline to Day 4 in log10 Hepatitis C Virus (HCV) RNA in Participants Without Baseline Drug Resistance
Description: The Roche TaqMan HCV quantitative assay was used for analysis with detection limit of 10 IU/mL. Baseline was Day -1.
Time Frame: Baseline to Day 4
Population: All randomized participants who took at least 1 dose of study medication and did not have baseline genotypic drug resistance mutations.
Measure: Mean (90% Confidence Interval); unit: log10 IU/mL
Arm/Group | Daclatasvir (1 mg) QD | Daclatasvir (10 mg) QD | Daclatasvir (30 mg) QD | Daclatasvir (60 mg) QD | Daclatasvir (30 mg) BID | Daclatasvir (100 mg) QD | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 3 | 3 | 3 | 6
log10 IU/mL | -2.16 [-2.68 to -1.64] | -3.29 [-3.81 to -2.77] | -3.04 [-3.56 to -2.52] | -3.85 [-4.45 to -3.25] | -3.82 [-4.42 to -3.22] | -3.14 [-3.74 to -2.54] | -0.07 [-0.49 to 0.36]

5. Secondary Outcome: Change From Baseline to Day 14 in Log10 Hepatitis C Virus (HCV) RNA in Participants Without Baseline Drug Resistance
Description: The Roche TaqMan HCV quantitative assay was used for analysis with detection limit of 10 IU/mL. Baseline was Day -1.
Time Frame: Baseline to Day 14
Population: as for outcome 4
Measure: Mean (90% Confidence Interval); unit: log10 IU/mL
Arm/Group | Daclatasvir (1 mg) QD | Daclatasvir (10 mg) QD | Daclatasvir (30 mg) QD | Daclatasvir (60 mg) QD | Daclatasvir (30 mg) BID | Daclatasvir (100 mg) QD | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 3 | 3 | 3 | 6
log10 IU/mL | -1.89 [-3.38 to -0.39] | -2.32 [-3.81 to -0.82] | -1.68 [-3.17 to -0.18] | -1.34 [-3.07 to 0.39] | -3.55 [-5.27 to -1.82] | -1.35 [-3.07 to 0.38] | -0.59 [-1.81 to 0.63]

6. Secondary Outcome: Time to Maximum Decline From Baseline in Hepatitis C Virus (HCV) RNA in Participants Without Baseline Drug Resistance
Description: Participants without baseline drug resistance were assessed for time to reach maximum decrease in log10 HCV RNA level.
Time Frame: Day 1 up to Day 14
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Daclatasvir (1 mg) QD | Daclatasvir (10 mg) QD | Daclatasvir (30 mg) QD | Daclatasvir (60 mg) QD | Daclatasvir (30 mg) BID | Daclatasvir (100 mg) QD | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 3 | 3 | 3 | 6
Days | 4.50 (4.726) | 5.25 (2.363) | 3.50 (2.380) | 3.33 (1.528) | 10.33 (6.028) | 7.67 (6.429) | 10.17 (6.524)

7. Secondary Outcome: Maximum Decline From Baseline in Log10 Hepatitis C Virus (HCV) RNA in Participants Without Baseline Drug Resistance
Description: The Roche TaqMan HCV quantitative assay was used for analysis with detection limit of 10 IU/mL.
Time Frame: Day 1 up to Day 14
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | Daclatasvir (1 mg) QD | Daclatasvir (10 mg) QD | Daclatasvir (30 mg) QD | Daclatasvir (60 mg) QD | Daclatasvir (30 mg) BID | Daclatasvir (100 mg) QD | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 3 | 3 | 3 | 6
log10 IU/mL | -2.81 (0.700) | -3.63 (0.776) | -3.31 (0.050) | -4.03 (0.626) | -4.88 (1.335) | -3.62 (0.170) | -1.32 (1.629)

8. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) and Minimum Observed Plasma Concentration (Cmin) of Daclatasvir on Days 1 and 14
Description: The peak concentrations in plasma (Cmax) and minimum observed plasma concentration (Cmin) were defined as the peak maximum and minimum plasma level of daclatasvir, derived from plasma concentration-time data analyzed by non-compartmental methods. Cmax and Cmin of daclatasvir in plasma was assayed using a validated liquid chromatography tandem mass spectrometry method.
Time Frame: 0 hour (pre-dose) 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 12 hours (post morning dose) at Day1 and Day 14, 0 hour (pre-dose) at Days 2, 3, 4, 5, 7, 9, 11, 13 and 24, 48 and 72 hours (post morning dose) at Day 14
Population: All participants who received at least 1 dose of study medication and with available Pharmacokinetic (PK) data were summarized.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliters(ng/mL)
Arm/Group | Daclatasvir (1 mg) QD | Daclatasvir (10 mg) QD | Daclatasvir (30 mg) QD | Daclatasvir (60 mg) QD | Daclatasvir (30 mg) BID | Daclatasvir (100 mg) QD
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4
nanograms/milliliters(ng/mL)
  Cmax at Day 1 | 15.731 (48) | 159.665 (41) | 483.365 (25) | 1409.202 (13) | 563.569 (26) | 1960.732 (21)
  Cmax at Day 14 | 10.430 (76) | 154.196 (49) | 555.878 (38) | 1726.383 (21) | 831.792 (37) | 1853.925 (26)
  Cmin at Day 1 | 1.212 (105) | 15.141 (49) | 41.114 (34) | 129.822 (25) | 171.330 (53) | 174.642 (21)
  Cmin at Day 14 | 1.234 (95) | 23.674 (53) | 61.635 (42) | 254.602 (42) | 206.941 (74) | 287.852 (37)

9. Secondary Outcome: Area Under the Concentration-time Curve (AUC) in 1 Dosing Interval of Daclatasvir at Days 1 and 14
Description: The area under the concentration-time curve in 1 Dosing Interval AUC(TAU) was used to measure the drug exposure over 1 dosing interval., derived from plasma concentration-time data analyzed by non-compartmental methods. AUC(TAU) of daclatasvir in plasma was assayed using a validated liquid chromatography tandem mass spectrometry method.
Time Frame: 0 hour (pre-dose) 0.5, 1,1.5, 2, 3, 4, 6, 8 and 12 hours (post morning dose) at Day1 and Day 14, 0 hr (pre-dose) at Days 2, 3, 4, 5, 7, 9, 11, 13, and 24, 48 and 72 hours (post morning dose) at Day 14
Population: All participants who received at least 1 dose of study medication and with available PK data were summarized.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Daclatasvir (1 mg) QD | Daclatasvir (10 mg) QD | Daclatasvir (30 mg) QD | Daclatasvir (60 mg) QD | Daclatasvir (30 mg) BID | Daclatasvir (100 mg) QD
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4
ng*h/mL
  Day 1 | 111.8 (54) | 1113.6 (38) | 3528.6 (19) | 10691.5 (20) | 3307.2 (36) | 15136.1 (19)
  Day 14 | 92.0 (80) | 1332.1 (46) | 4391.3 (27) | 15120.9 (35) | 5431.6 (35) | 17592.8 (15)

10. Secondary Outcome: Plasma Half-life (T-half) of Daclatasvir at Day 14
Description: The absolute values of lamda (λ) were used to evaluate apparent terminal half-life (T-half) was defined as T-half= ln 2/λ. T-half was derived from plasma concentration-time data analyzed by non-compartmental methods. T-half of daclatasvir in plasma was assayed using a validated liquid chromatography tandem mass spectrometry method.
Time Frame: as for outcome 9
Population: All participants who received at least 1 dose of study medication and with available PK data were summarized.
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Daclatasvir (1 mg) QD | Daclatasvir (10 mg) QD | Daclatasvir (30 mg) QD | Daclatasvir (60 mg) QD | Daclatasvir (30 mg) BID | Daclatasvir (100 mg) QD
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4
h | 11.68 (2.214) | 14.31 (3.848) | 12.99 (2.039) | 12.81 (1.233) | 13.04 (3.654) | 15.19 (3.411)

11. Secondary Outcome: Apparent Total Body Clearance (CLT/F) of Daclatasvir on Day 14
Description: The apparent total body clearance at steady state (CLT/F) was defined as the apparent body clearance of canakinumab from the serum when the systemic availability was unknown. CLT/F was derived from plasma concentration-time data analyzed by non-compartmental methods. CLT/F of daclatasvir in plasma was assayed using a validated liquid chromatography tandem mass spectrometry method.
Time Frame: 0 hour (pre-dose) 0.5, 1,1.5, 2, 3, 4, 6, 8 and 12 hours (post morning dose) at Day1 and Day 14, 0 hour (pre-dose) at Days 2, 3, 4, 5, 7, 9, 11, 13, and 24, 48 and 72 hours (post morning dose) at Day 14
Population: All participants who received at least 1 dose of study medication and with available PK data were summarized.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | Daclatasvir (1 mg) QD | Daclatasvir (10 mg) QD | Daclatasvir (30 mg) QD | Daclatasvir (60 mg) QD | Daclatasvir (30 mg) BID | Daclatasvir (100 mg) QD
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4
mL/min | 181.118 (52) | 125.119 (52) | 113.861 (25) | 66.133 (29) | 92.054 (35) | 94.736 (15)

12. Secondary Outcome: Average Observed Plasma Concentration (Css-av) at Steady State of Daclatasvir at Days 1 and 14
Description: The average observed plasma concentration at steady state (Css-av) was calculated as ratio of AUC(TAU) by TAU, where TAU = 24 h for QD dosing and 12 h for BID dosing. Css-av was derived from plasma concentration-time data analyzed by non-compartmental methods. Css-av of daclatasvir in plasma was assayed using a validated liquid chromatography tandem mass spectrometry method.
Time Frame: 0 hour (pre-dose) 0.5, 1,1.5, 2, 3, 4, 6, 8 and 12 hours (post morning dose) at Day1 and Day 14, 0 hr (pre-dose) at Days 2, 3, 4, 5, 7, 9, 11,13, and 24, 48 and 72 hours (post morning dose) at Day 14
Population: All participants who received at least 1 dose of study medication and with available PK data were summarized.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Daclatasvir (1 mg) QD | Daclatasvir (10 mg) QD | Daclatasvir (30 mg) QD | Daclatasvir (60 mg) QD | Daclatasvir (30 mg) BID | Daclatasvir (100 mg) QD
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4
ng/mL
  Day 1 | 4.659 (54) | 46.401 (38) | 147.024 (19) | 445.478 (20) | 275.596 (36) | 630.673 (19)
  Day 14 | 3.834 (80) | 55.503 (46) | 182.972 (27) | 630.039 (35) | 452.634 (35) | 733.035 (15)

13. Secondary Outcome: Accumulation Index (AI) AUC(TAU), AI Cmax, and Degree of Fluctuation (DF) of Daclatasvir on Day 14
Description: Accumulation index area under the concentration-time curve of daclatasvir to the end of the dosing period [AI AUC(TAU)] was defined as the ratio of AUC(TAU) at steady-state to AUC(TAU) after the first dose.Accumulation index maximum observed concentration of daclatasvir in plasma (AI Cmax) was defined as the ratio of Cmax at steady-state to Cmax after the first dose. Degree of Fluctuation (DF) was defined as the ratio of difference between Cmax and Cmin at steady state by Css-av. The parameters were analyzed using non-compartmental methods, assayed by validated liquid chromatography tandem mass spectrometry (LC-MS/MS).
Time Frame: as for outcome 11
Population: All participants who received at least 1 dose of study medication and with available PK data were summarized.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Daclatasvir (1 mg) QD | Daclatasvir (10 mg) QD | Daclatasvir (30 mg) QD | Daclatasvir (60 mg) QD | Daclatasvir (30 mg) BID | Daclatasvir (100 mg) QD
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4
ratio
  AI AUC(TAU) | 0.823 (29) | 1.196 (16) | 1.245 (20) | 1.414 (17) | 1.642 (16) | 1.162 (25)
  AI Cmax | 0.663 (57) | 0.966 (26) | 1.150 (28) | 1.225 (10) | 1.476 (32) | 0.946 (42)
  Degree of Fluctuation | 2.389 (13) | 2.335 (18) | 2.659 (25) | 2.321 (24) | 1.251 (18) | 2.133 (12)

14. Secondary Outcome: Time of Maximum Observed Plasma Concentration (Tmax) of Daclatasvir on Days 1 and 14
Description: Tmax was defined as the time to reach maximum observed plasma concentration of daclatasvir in plasma. Tmax was derived from plasma concentration-time data analyzed by non-compartmental methods. Tmax of daclatasvir in plasma was assayed using a validated liquid chromatography tandem mass spectrometry method.
Time Frame: as for outcome 11
Population: All participants who received at least 1 dose of study medication and with available PK data were summarized.
Measure: Median (Full Range); unit: h
Arm/Group | Daclatasvir (1 mg) QD | Daclatasvir (10 mg) QD | Daclatasvir (30 mg) QD | Daclatasvir (60 mg) QD | Daclatasvir (30 mg) BID | Daclatasvir (100 mg) QD
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4
h
  Day 1 | 2.000 [1.00 to 3.00] | 1.000 [1.00 to 2.00] | 1.000 [0.50 to 1.00] | 1.500 [1.50 to 3.00] | 2.500 [1.50 to 3.00] | 1.500 [1.00 to 1.50]
  Day 14 | 1.250 [1.00 to 2.00] | 1.250 [1.00 to 1.50] | 1.000 [1.00 to 1.50] | 1.000 [1.00 to 2.00] | 1.750 [1.00 to 2.00] | 1.750 [1.00 to 2.00]

15. Secondary Outcome: Correlation Coefficients Between Measures of Decline in log10 Hepatitis C Virus (HCV) RNA and Daclatasvir PK Parameters Cmax, AUC(TAU), and Cmin on Day 14 in Participants Without Baseline Drug Resistance
Description: Correlation between decline of log10 hepatitis C virus (HCV) RNA and exposure to study drug was measured by Pearson Correlation Coefficients. The change from baseline at Day 4 in log10 HCV RNA and the maximum decline in log10 HCV RNA were evaluated against the PK parameters Cmax, Cmin and AUC(TAU).
Time Frame: Day 4, Day 14
Population: All participants who received at least 1 dose of daclatasvir and who had no baseline genotype resistance were analyzed. Placebo participants were excluded from this analysis.
Measure: Number; unit: Correlation Coefficient
Groups:
- All Daclatasvir Treated Participants: All participants who received daclatasvir during 14 day treatment period.
Arm/Group | All Daclatasvir Treated Participants
Number analyzed (Participants) | 21
Correlation Coefficient
  Cmax and Delta log10 HCV RNA at Day 4 | -0.61
  AUC(Tau) and Delta log10 HCV RNA at Day 4 | -0.61
  Cmin and Delta log10 HCV RNA at Day 4 | -0.63
  Cmax and Maximum Decline in log10 HCV RNA | -0.51
  AUC(Tau) and Maximum Decline in log10 HCV RNA | -0.50
  Cmin and Maximum Decline in log10 HCV RNA | -0.59

16. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs), Discontinuation Due to Adverse Events (AEs), and Who Died
Description: AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization.
Time Frame: Day 1 to Day 182 or Day of Discharge
Population: All participants who received study drug were summarized.
Measure: Number; unit: participants
Arm/Group | Daclatasvir (1 mg) QD | Daclatasvir (10 mg) QD | Daclatasvir (30 mg) QD | Daclatasvir (60 mg) QD | Daclatasvir (30 mg) BID | Daclatasvir (100 mg) QD | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 6
participants
  SAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Discontinuation Due to AEs | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Death | 0 | 0 | 0 | 0 | 0 | 0 | 0

17. Secondary Outcome: Number of Participants With Marked Laboratory Abnormalities in Hematology
Description: Hematology marked laboratory abnormalities were defined as Hemoglobin (g/dL) Low as < 0.85*Pre-therapy (PreRx), Hematocrit (%) Low as < 0.85*PreRx, Platelet Count *10^9 c/L Low as < 0.85*Lower Limits of Normal (LLN) if PreRx = Missing/< 0.85*LLN if PreRx >= LLN/< 0.85*PreRx if PreRx < LLN, Eosinophils (absolute) *10^3 c/µL High as > 0.75*count, Leukocytes White Blood Cell (WBC) *10^3 c/µL High as > 1.2*ULN if LLN <= PreRx <= Upper Limits of Normal (ULN) > 1.2*ULN if PreRx = Missing/> 1.5*PreRx if PreRx > ULN/> ULN if PreRx < LLN.
Time Frame: Screening, Day 3, Day 7, Day 11, Day 14, and Day 28
Population: All participants treated with study drug were summarized.
Measure: Number; unit: participants
Arm/Group | Daclatasvir (1 mg) QD | Daclatasvir (10 mg) QD | Daclatasvir (30 mg) QD | Daclatasvir (60 mg) QD | Daclatasvir (30 mg) BID | Daclatasvir (100 mg) QD | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 6
participants
  Low Hematocrit | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Low Hemoglobin | 1 | 0 | 0 | 1 | 0 | 0 | 1
  Low Platelet | 0 | 0 | 0 | 0 | 0 | 1 | 0
  High Eosinophils | 0 | 0 | 0 | 0 | 0 | 1 | 0
  High Leukocytes | 0 | 0 | 0 | 0 | 0 | 1 | 0

18. Secondary Outcome: Number of Participants With Marked Abnormalities in Liver and Kidney Function Laboratory Tests and Electrolytes
Description: Liver and kidney function marked laboratory abnormalities were defined as Alanine Aminotransferase (ALT) units per liter (U/L) High as > 1.25*PreRx if PreRx > ULN/> 1.25*ULN if PreRx <= ULN/> 1.25*ULN if PreRx = Missing, Aspartate Aminotransferase (AST) U/L High as > 1.25* PreRx if PreRx > ULN/> 1.25*ULN if PreRx <= ULN/> 1.25*ULN if PreRx = Missing, Alkaline Phosphatase(ALP)U/L High as > 1.25*PreRx if PreRx > ULN/> 1.25*ULN if PreRx <= ULN/> 1.25*ULN if PreRx = Missing, G-Glutamyl Transferase (GGT) in U/L High as >1.15*ULN if PreRx<=ULN/>1.15* if PreRx missing/>1.2* PreRx if PreRx>ULN, Phosphorus Inorganic (mg/dL) Low as < 0.85*LLN if LLN <= PreRx <= ULN/< 0.85*LLN if PreRx = Missing/< 0.85*PreRx if PreRx < LLN/< LLN if PreRx > ULN, and Potassium serum milliequivalents per liter (mEq/L) High as > 1.1*PreRx if PreRx > ULN/> 1.1*ULN if LLN <= PreRx <= ULN/> 1.1*ULN if PreRx = Missing/> ULN if PreRx < LLN.
Time Frame: Screening, Day 3, Day 7, Day 11, Day 14, and Day 28
Population: All participants who were treated with study drug were summarized.
Measure: Number; unit: participants
Arm/Group | Daclatasvir (1 mg) QD | Daclatasvir (10 mg) QD | Daclatasvir (30 mg) QD | Daclatasvir (60 mg) QD | Daclatasvir (30 mg) BID | Daclatasvir (100 mg) QD | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 6
participants
  ALT High | 0 | 1 | 0 | 1 | 2 | 2 | 0
  AST High | 0 | 1 | 0 | 0 | 2 | 2 | 1
  ALP High | 0 | 0 | 0 | 0 | 0 | 1 | 0
  GGT | 0 | 0 | 2 | 0 | 2 | 1 | 2
  Phosporus Low | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Potassium High | 0 | 0 | 1 | 0 | 0 | 0 | 1

19. Secondary Outcome: Number of Participants With Marked Laboratory Abnormalities in Lipase and Glucose
Description: Marked abnormalities were defined as Lipase (U/L) High as >1.5*ULN, Glucose fasting serum (mg/dL) High as > 1.3*ULN if LLN <= PreRx <= ULN/> 1.3*ULN if PreRx = Missing/>2*PreRx; if PreRx > ULN/> ULN if PreRx < LLN.
Time Frame: Screening, Day 3, Day 7, Day 11, Day 14, and Day 28
Population: All participants treated with study drug were summarized.
Measure: Number; unit: participants
Arm/Group | Daclatasvir (1 mg) QD | Daclatasvir (10 mg) QD | Daclatasvir (30 mg) QD | Daclatasvir (60 mg) QD | Daclatasvir (30 mg) BID | Daclatasvir (100 mg) QD | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 6
participants
  Lipase High | 0 | 1 | 0 | 0 | 1 | 0 | 0
  Glucose Fasting High | 0 | 0 | 0 | 0 | 0 | 1 | 1

20. Secondary Outcome: Number of Participants With Marked Laboratory Abnormalities in Urinalysis
Description: Marked laboratory abnormalities in urinalysis were defined as, Blood Urine High as >= 2*PreRx if PreRx >= 1/>= 2 if PreRx < 1/>= 2 if PreRx = Missing. Glucose Urine High as >= 1 if PreRx < 1/>= 1 if PreRx = Missing/>= 2*PreRx if PreRx >= 1.
Time Frame: Screening, Day 3, Day 7, Day 11, Day 14, and Day 28
Population: All participants treated with study drug were summarized.
Measure: Number; unit: participants
Arm/Group | Daclatasvir (1 mg) QD | Daclatasvir (10 mg) QD | Daclatasvir (30 mg) QD | Daclatasvir (60 mg) QD | Daclatasvir (30 mg) BID | Daclatasvir (100 mg) QD | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 6
participants
  Urine Blood High | 1 | 1 | 0 | 1 | 0 | 0 | 1
  Urine Glucose High | 1 | 0 | 0 | 0 | 0 | 0 | 2

21. Secondary Outcome: Number of Participants With Clinically Relevant Change From Baseline in Vital Signs
Description: Vital signs included: body temperature, respiratory rate, blood pressure (systolic and diastolic) and heart rate. Blood pressure and heart rate were measured after the participant had been supine, semi-supine, or seated quietly for at least 5 minutes. Baseline was defined as the last observation prior to dosing on Day 1.
Time Frame: Screening, Day -1 and prior to morning dose on Day 1, 2, 14, and 28
Population: All participants treated with study drug were summarized.
Measure: Number; unit: participants
Arm/Group | Daclatasvir (1 mg) QD | Daclatasvir (10 mg) QD | Daclatasvir (30 mg) QD | Daclatasvir (60 mg) QD | Daclatasvir (30 mg) BID | Daclatasvir (100 mg) QD | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 6
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

22. Secondary Outcome: Number of Participants Meeting Pre-Specified Criteria in Electrocardiogram Parameters
Description: Pre-specified criteria were defined as, Heart rate (HR) minimum as <=50 bpm/change from baseline <-20 bpm/maximum HR >100 bpm, QT interval corrected using Fridericia's formula (QTcF) maximum as QTcF<=450 msec/450 msec <maximum QTcF and <=480 msec/480 msec <maximum QTcF <= 500 msec/maximum QTcF>500 msec, QRS interval as <=120 msec/>120 msec, and PR interval maximum as <= 200 msec/>200 msec.
Time Frame: Screening, Day 2, 3, 5, 7, 9, 11, 13, 15, 21 and 28
Population: All participants treated with study drug were summarized.
Measure: Number; unit: participants
Arm/Group | Daclatasvir (1 mg) QD | Daclatasvir (10 mg) QD | Daclatasvir (30 mg) QD | Daclatasvir (60 mg) QD | Daclatasvir (30 mg) BID | Daclatasvir (100 mg) QD | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 6
participants
  Heart Rate <=50 bpm | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Heart Rate > 100 bpm | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HR Change from baseline <-20bpm | 0 | 0 | 0 | 0 | 4 | 0 | 0
  Maximum QTcF <= 450 msec | 4 | 4 | 4 | 4 | 4 | 4 | 6
  Maximum QTcF >450 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Maximum Delta QTcF<=30 | 4 | 4 | 4 | 4 | 4 | 4 | 6
  Maximum Delta QTcF >30 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Maximum QRS <=120 msec | 4 | 4 | 4 | 4 | 4 | 4 | 6
  Maximum QRS > 120 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Maximum PR <=200 msec | 4 | 4 | 4 | 4 | 4 | 4 | 6
  Maximum PR > 200 msec | 0 | 0 | 0 | 0 | 0 | 1 | 0

ADVERSE EVENTS:
Arm/Group | Daclatasvir (1 mg) QD | Daclatasvir (10 mg) QD | Daclatasvir (100 mg) QD | Daclatasvir (30 mg) BID | Daclatasvir (30 mg) QD | Daclatasvir (60 mg) QD | Placebo
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/4 | 0/4 | 0/4 | 0/6
Other Adverse Events (participants affected / at risk) | 1/4 | 4/4 | 2/4 | 2/4 | 3/4 | 4/4 | 4/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Daclatasvir (1 mg) QD (N=4) | Daclatasvir (10 mg) QD (N=4) | Daclatasvir (100 mg) QD (N=4) | Daclatasvir (30 mg) BID (N=4) | Daclatasvir (30 mg) QD (N=4) | Daclatasvir (60 mg) QD (N=4) | Placebo (N=6)
Eye injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urethritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 1 | 1 | 0 | 2 | 2
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Restlessness (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Visual acuity reduced (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Energy increased (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Electrocardiogram T wave abnormal (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Faeces discoloured (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nightmare (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinus headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sleep disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tongue injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.